CLINICAL TRIAL: NCT00877097
Title: Randomized Clinical Trial on the Effectts of Estradiol 2 mg + NETA 1 mg With or Without Clodronate on Bone Mineral Density and Bone Markers of Osteoporotic Postmenopausal 167 Finnish Women.
Brief Title: Effects of Continuous Combined Hormone Replacement Therapy and Clodronate on Bone Mineral Density (BMD) in Osteoporotic Women
Acronym: Osteo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Mari Ollikainen, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUH5302410; Compliance 1x/year x5; BP 1x/year 5 yrs; endometrial sample 1x/yearx5; adverse effects 1x/year x5
Record Dates: First submitted 2009-04-02; First posted 2009-04-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Osteoporosis
Keywords: osteoporosis; Bone mineral density; clodronate; HRT; postmenopausal
MeSH Terms: conditions — Osteoporosis | interventions — Trisequens; Clodronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Clodronate 800 mg / day + estradiol 2 mg + norethisterone acetate 1 mg / day for five years.
  Interventions: Drug: Klodronate and Kliogest
- 2 (Placebo Comparator): Placebo 2 tablets/ day + estradiol 2 mg + norethisterone acetate 1 mg / day for five years.
  Interventions: Procedure: Placebo+ Kliogest
- 3 (Active Comparator): Clodronate 800 mg / day for five years.
  Interventions: Drug: Bonefos

INTERVENTIONS:
Drug: Klodronate and Kliogest
  Arms: 1
Procedure: Placebo+ Kliogest
  Arms: 2
Drug: Bonefos
  Arms: 3

SUMMARY:
Recent studies suggest that the combination of two inhibitors of bone resorption may induce a greater increase in bone mineral density (BMD) than either agent alone.

In this 5-year partly randomized study the investigators examined the effects of hormone therapy (HT) with or without bisphosphonate on BMD on osteoporotic women.

In the Kuopio Osteoporosis Study (OSTPRE) a population based sample of 3200 women were selected for BMD measurement by Lunar DPX in 1995-1997. In all 167 women aged 61±2.7 years (11±4.9 years postmenopausal), and the T-score < -2.5 SD at either the lumbar spine or femoral neck were recruited for this sub-study.

They received daily estradiol hemihydrate (E2) 2mg + norethisterone acetate (NETA) 1mg (Kliogest®, Novo Nordisk, Denmark) and were randomized to get additional Boneplac, which consisted of either 800mg clodronate (Bonefos®, Leiras Ltd, Finland) (n=55, KB-group) or placebo (n=55, K-group). In case of contraindications or refusal from HT, the women were offered clodronate 800 mg/day (n=57, B-group) to be taken to empty stomach with a glass of water 30 minutes to two hours before breakfast.

BMD was measured at time intervals 0, 1, 3 and 5-years. All repeated BMD values were interviewed by one investigator and primarily the vertebrae L2-L4 were followed. In case of spinal deformities during the study (38.3%) other lumbar levels were followed. The baseline BMD values (lumbar spine BMD 0.839±0.072 g/cm², femoral neck BMD 0.759±0.094g/cm²) were similar between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* BMD T-score <-2.5sd

Exclusion Criteria:

* None

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 1996-07; Primary Completion 2002-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
BMD once a year | 1996-2002

SECONDARY OUTCOMES:
bone markers once a year | 1996-2002

CONTACTS AND LOCATIONS:
Overall Officials: Marjo T Tuppurainen, MD, PhD, Principal Investigator — Dept. of Obstetrics and Gynecology, Kuopio University Hospital

REFERENCES:
- [Derived] Tuppurainen M, Harma K, Komulainen M, Kiviniemi V, Kroger H, Honkanen R, Alhava E, Jurvelin J, Saarikoski S. Effects of continuous combined hormone replacement therapy and clodronate on bone mineral density in osteoporotic postmenopausal women: a 5-year follow-up. Maturitas. 2010 Aug;66(4):423-30. doi: 10.1016/j.maturitas.2010.04.013. Epub 2010 May 23. PMID 20547017